CLINICAL TRIAL: NCT03686202
Title: Feasibility Study of Microbial Ecosystem Therapeutics (MET-4) to Evaluate Effects of Fecal Microbiome in Patients on ImmunOtherapy (MET4-IO)
Brief Title: Feasibility Study of MET-4: Evaluating Fecal Microbiome Effects in Immunotherapy Patients
Acronym: MET4-IO
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MET4-IO-001
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: All Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Safety Cohort (Experimental): Subjects with advanced solid tumors already on ICI will receive treatment with MET-4 in addition to SOC ICI. MET-4 is administered orally as an initial daily loading dose (5g) of MET-4 over 2 days followed by a daily maintenance dose (1.5g) of MET-4 and will be continued until unacceptable toxicity, progression of disease
  Interventions: Biological: MET-4
- Group B (Experimental): Eligible subjects with advanced solid tumors starting ICI will be randomised in a 3:1 ratio stratifying for prior IO exposure, to receive MET-4 together with any approved PD-1/PD-L1 inhibitor as per SOC or control group. There will be a run-in period for subjects in the MET-4 treatment group. Following the run-in period of ICI therapy, subjects will be administered the same MET-4 dose as subjects in group A.
  Interventions: Biological: MET-4
- Group C (Experimental): In group C, eligible subjects with advanced solid tumors whom are already on ICI with first unconfirmed PD on evaluation scans per investigator's assessment, will be randomised in a 1:1 ratio to receive MET-4 in addition to the PD-1/PD-L1 inhibitor as per SOC or control group. These subjects must be clinically stable and are to be continued on ICI at the discretion of the investigator. There will be no run-in period for this cohort. Subjects will be administered the same MET-4 dose as subjects in groups A and B.
  Interventions: Biological: MET-4
- Group D (Experimental): In group D, eligible subjects with stage III or resected stage IV melanoma who are to start adjuvant ICI, will be randomized in a 1:1 ratio to receive MET-4 in addition to anti-PD1 antibody +/- anti-CTLA4 antibody as per SOC or control group. Patients will be stratified per BRAF mutation status. Subjects will be administered the same MET-4 dose as subjects in groups A, B and C. MET-4 will be initiated as run-in for a minimum of 1 week, and maximum of 2 weeks before ICI administration. MET-4 will be continued until unacceptable toxicity, confirmed PD by RECIST v1.1 or completion of 1 year of ICI, whichever occurs earlier. Subjects in the control arms of groups B, C and D will be treated with ICI therapy as per institution standard of care without MET-4.
  Interventions: Biological: MET-4

INTERVENTIONS:
Biological: MET-4 — Microbial Ecosystem Therapeutics (MET) is a new treatment approach developed as an alternative to fecal transplantation. Unlike donor stool used in fecal transplants, which are incompletely characterised complex communities of microbes and associated metabolites and fecal material, MET consists of a defined mixture of pure live cultures of intestinal bacteria isolated from a stool sample of a healthy donor.

SUMMARY:
This study is designed to assess the safety, tolerability and engraftment (cumulative relative abundance) of MET-4 strains when given in combination with immune checkpoint inhibitors (ICIs). There will be a safety cohort (group A) of 5 subjects which will receive MET-4 in addition to standard of care (SOC) ICI. After the safety cohort, 40 patients will be enrolled in group B which will be randomized to MET4 with SOC ICI vs. control group with SOC ICI only. Group C will enroll 20 patients who have already started on SOC ICI and have had first unconfirmed progression of disease and expected to continue with standard ICI treatment. These patients will be randomized to continue receiving standard ICI alone, or SOC ICI with MET4.

DETAILED DESCRIPTION:
Human associated microorganisms (the microbiota) inhabit virtually all surfaces of the human body. The gut is densely colonized by the microbiota which aids in the digestion. Animal and human observational and experimental evidence show a link between gut microbiota and the activation, regulation and function of the immune system. Pre-clinical studies in mouse models have linked the gut microbiota to efficacy of anticancer therapies. Microbial Ecosystem Therapeutics (MET) is a new treatment approach developed as an alternative to fecal transplantation. MET consists of a defined mixture of pure live cultures of intestinal bacteria isolated from a stool sample of a healthy donor.

This study is designed to assess the safety, tolerability and engraftment (cumulative relative abundance) of MET-4 strains when given in combination with immune checkpoint inhibitors (ICIs).

ELIGIBILITY:
Inclusion Criteria:

* Signed written and voluntary informed consent
* Age >=18 years, male or female
* Histologically or cytological documented locally-advanced or metastatic solid malignancy which is incurable.
* Group A: Is already on treatment with monotherapy anti-PD-1 or PD-L1 immune checkpoint inhibitor, not in the context of a therapeutic clinical trial.

Group B: Is intended to start on treatment with monotherapy anti-PD-1 or PD-L1 immune checkpoint inhibitors as considered appropriate by treatment physician, and not in the context of a therapeutic clinical trial.

Group C: Is already on treatment with monotherapy anti-PD-1 or PD-L1 immune checkpoint inhibitor, not in the context of a therapeutic clinical trial with first unconfirmed PD on evaluation scan per investigator's assessment.

* Be willing to provide 10-15 unstained slides of archival tissue sample. Subjects who decline or have not sufficient archived tissue samples may still enroll if all other criteria are eligible.
* Be willing and able to provide stool and blood specimen for analyses at protocol specified time points.
* Have measurable disease based on RECIST 1.1
* Performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Prior therapy with any immunotherapy allowed.
* Not pregnant for females of child bearing potential as indicated by negative serum or urine pregnancy test within 72 hours of study start.

Exclusion Criteria:

* Subjects unable to swallow orally administered medications or any subjects with gastrointestinal disorders likely to interfere with absorption (e.g. bowel obstruction, short gut syndrome, blind loop syndrome, ileostomy etc). Subjects with colostomies may be enrolled.
* Any condition that, in the opinion of the Investigator, would interfere with subject safety, or evaluation of the collected specimen and interpretation of study result.
* Pregnant or planning to get pregnant in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative relative abundance of immunotherapy-responsiveness associated species at day 12 of MET-4 | Approximately 12 days
  Fecal microbial abundance measured via qPCR and Nanostring analysis of stool at approximately day 12
Changes in relative abundance of immunotherapy-responsiveness associated MET-4 strains between baseline and approximately day 12 | Approximately 12 days
  Microbiome gene sequencing of stool at baseline and approximately day 12 post first dose
Number of participants with treatment-related adverse events assessed by CTCAE v.5.0 | 2 years
  Related toxicities and severity collected as per CTCAE version 5.0

SECONDARY OUTCOMES:
Cumulative relative abundance of immunotherapy-responsiveness associated species at later MET-4 or control time points (approximately 24 weeks and/or 1-2 weeks following the end of treatment). | 2 years
  Fecal microbial abundance measured via qPCR and Nanostring analysis of stool at baseline and week 24 after first dose and EOT.
Changes in relative abundance of immunotherapy-responsiveness associated MET-4 strains between baseline and later MET-4 or control timepoints (approximately 24 weeks and/or 1-2 weeks following the end of treatment) | 2 years
  Microbiome gene sequencing of stool at baseline and week 24 after first dose and EOT.
Bacterial taxonomic diversity between baseline and follow-up samples | 2 years
  Microbiome gene sequencing of stool at baseline, day 10-16 post first dose, week 3-4 post first dose, and week 24 after first dose and EOT.

OTHER OUTCOMES:
Response | 2 years
  Objective response rates of ICI when given in combination with MET-4 as measured per RECIST v1.1 and iRECIST
Progression free survival | 2 years
  Time from randomization until disease progression or death as measured per RECIST v.1.1 and iRECIST
Changes in immune cell subsets in the systemic circulation in response to MET-4 through serial blood sampling. | 24 weeks
  Flow cytometry/CyTOF of blood at baseline, 6-8 weeks post first dose of MET, 24 weeks post first dose
Characterization of tumor microenvironment of archived tumor samples | 2 years
  Standard immunohistochemistry (IHC) of baseline archival tumor
Dynamic measures of microbiome as correlates of blood immune profiling | 2 years
  Flow cytometry/CyTOF of blood at baseline, week 3-4 post first dose of MET, and week 24 post first dose, and stool microbiome gene profiling at baseline, 10-16 days first dose of MET, week 3-4 post first dose, week 24 post first dose and end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre; Anna Spreafico, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No